CLINICAL TRIAL: NCT00865722
Title: Pilot Study to Test Feasibility, Safety, Molecular Mediators and Preliminary Efficacy of Remote Myocardial Postconditioning Provided With Extrinsic Cuff Compression of Lower Limb During Primary PCI
Brief Title: Remote Postconditioning in Patients With Acute Myocardial Infarction Treated by Primary Percutaneous Coronary Intervention (PCI)
Acronym: RemPostCon
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Maurizio Ferrario, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RemPostConditioning
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Myocardial Reperfusion Injury; Myocardial Ischemia; Myocardial Infarction
Keywords: Remote Postconditioning; Myocardial reperfusion Injury; Myocardial Infarction; Primary PCI
MeSH Terms: conditions — Myocardial Reperfusion Injury; Myocardial Ischemia; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RemotePostConditioning (Active Comparator): Patients will receive pPCI and treatments according to guidelines for STEMI PLUS extrinsic cuff compression to the lower limb for 5 ' followed by 5' reperfusion for three cycles (30' in total) starting with myocardial reperfusion
  Interventions: Procedure: Remote Postconditioning
- Controls (Sham Comparator): pPCI and treatments according to guidelines for STEMI
  Interventions: Procedure: Remote Postconditioning

INTERVENTIONS:
Procedure: Remote Postconditioning — Lower limb compression using a cuff inflated to 200 mmHg for 5 ' followed by 5' of reperfusion fo three times during 30'

SUMMARY:
Background: Experimental studies suggest that remote limb ischaemic postconditioning (RemPostCon) can reduce infarct size in pigs. Initial clinical applications support the beneficial role of RemPostCon in preserving endothelial function during upper limb ischemia in healthy volunteers and in patients with stable coronary artery disease.

Aim of the study: To evaluate the feasibility, safety and efficacy of RemPostCon in the setting of STEMI and primary PCI (pPCI) and to investigate potential circulating mediators of its effects.

Patients and methods: Patients who undergo pPCI for anterior STEMI within 6 hours since the onset of symptoms are randomly assigned to receive either RemPostCon + pPCI or pPCI alone in a single-blind fashion. All patients receive therapy according to the current international guidelines. Three cycles of ischemia-reperfusion are provided to the lower limb inflating a cuff to 200 mmHg. Each cycle consists of 5' of ischaemia, followed by 5' of reperfusion. RemPostCon is started at the time of angioplasty in the infarct related artery. Primary endpoint is the area under the curve (AUC) of creatinine kinase - MB (CK - MB). Cardiac magnetic resonance (CMR) is performed early before discharge and 4 months after the event, if there are no contraindications.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 yrs AND Age =< 80 yrs
* STEMI definition
* Pain to door time < 6 hrs
* Killip class 1 - 2 - 3
* Initial TIMI flow 0 - 1 in the anterior descending artery
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Cardiogenic shock
* Initial TIMI flow 2 - 3 in the anterior descending artery
* History of prior MI in the past 6 months
* History of prior CABG
* History of peripheral vascular disease III - IV grade
* History of abdominal Aortic Aneurysm > 5 cm
* Severe coronaropathy that could condition further revascularization before the end of the study
* Other relevant medical or surgical conditions that can influence prognosis at 4 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve of CK - MB release | baseline to 72h since admission

SECONDARY OUTCOMES:
Area Under the Curve of CK release | baselinte to 72h since admission
TIMI Frame Count | 30 minutes after first balloon inflation in infarct-related artery
Time to balloon | during pPCI
Ejection Fraction MRI | before discharge and after 4 months
Myocardial Blush grading | 30 minutes after first balloon inflation
ST segment resolution | 6h after balloon
Troponin I peak | 72h since admission
Mortality rate | 4 months since admission
artero-venous differences in pO2, pCO2, pH, HCo3 | baseline and 30 minutes after first balloon inflation
Major adverse cardiac events | 4 months since admission
artero-venous quantitative and qualitative differences in endothelial progenitors cells (subgroups) | within 24 h since admission
artero-venous Differences of Cytokines | within 24h since admission
Edema Volume T2 sequences MRI | before discharge
Delay enhancement volume MRI | before discharge and after 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Ferrario, MD, Study Director — IRCCS Policlinico San Matteo; Gabriele Crimi, MD, Principal Investigator — IRCCS Policlinico San Matteo
Locations (2):
- Italy (2):
  - IRCCS Policlinico San Matteo, Pavia, Italy
  - ASL3 Genovese, Villa Scassi Hospitale, Genoa

REFERENCES:
- [Derived] Crimi G, Pica S, Raineri C, Bramucci E, De Ferrari GM, Klersy C, Ferlini M, Marinoni B, Repetto A, Romeo M, Rosti V, Massa M, Raisaro A, Leonardi S, Rubartelli P, Oltrona Visconti L, Ferrario M. Remote ischemic post-conditioning of the lower limb during primary percutaneous coronary intervention safely reduces enzymatic infarct size in anterior myocardial infarction: a randomized controlled trial. JACC Cardiovasc Interv. 2013 Oct;6(10):1055-63. doi: 10.1016/j.jcin.2013.05.011. PMID 24156966